CLINICAL TRIAL: NCT02234505
Title: Physiologic Range of Step-by-step Variations in Lower Limb Prosthesis Forces
Brief Title: Physiologic Range of Step-by-step Variations in Lower Limb Prosthesis Forces During Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Orthotic and Prosthetic Association (Other)
Responsible Party: Principal Investigator, Goeran Fiedler, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO14040403
Record Dates: First submitted 2014-08-28; First posted 2014-09-09 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Trans-tibial Limb Loss
Keywords: prosthetics; amputation; gait stability; step variability; load cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trans-tibial prosthesis users (Experimental): prosthetic alignment perturbation
  Interventions: Procedure: Prosthetic alignment perturbation

INTERVENTIONS:
Procedure: Prosthetic alignment perturbation — Prosthetic ankle plantar-flexion will be modified in different degrees, devices (prosthetic components) will not be modified from baseline condition

SUMMARY:
In human gait there is a certain amount of variation between steps; some considered physiological and owed to variations in environment or posture, and some severe enough to be indicative of gait instabilities that may lead to stumbling and falling. In users of lower limb prosthetics, such gait instabilities are of especially great interest.

The study investigates the correlation between socket alignment quality and gait step-by-step variability in users of trans-tibial-prosthetics. It is hypothesized that a clearly defined range of step-by-step variability exists, and that therefore step-by-step variability is suitable as an outcome variable for the assessment of socket alignment.

A sample of ten persons with trans-tibial amputation will be recruited for this pilot study. Subjects will be asked to walk on different natural surfaces while the socket alignment is successively perturbed. Step-by-step variations in horizontal ground reaction forces and torsional moments will be measured and statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* activity classification of K2 to K4
* experience in prosthesis use of at least one year
* stated ability to walk pain free for at least 30 minutes

Exclusion Criteria:

* age of less than 18 years
* acute or ongoing residual limb pain
* use of a prosthesis that is not suitable for installation of the load cell (e.g. is too short, or has non-removable cosmesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Step-by-step variability | 2 hours
  Peak horizontal ground reaction force (Fx and Fy) as well as peak axial torsion moment (Mz) will be extracted for 10 consecutive intermediary steps for each testing condition. Total range in Newtons over the 10 step sample, as well as maximal difference between consecutive steps in Newtons and percent will be reported for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakery Square MSPO labs, Pittsburgh, Pennsylvania, United States